CLINICAL TRIAL: NCT01956643
Title: Effect of Sham Feeding on Postoperative Ileus After Elective Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ho Geol Ryu, Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ShamLT
Record Dates: First submitted 2013-09-27; First posted 2013-10-08 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Postoperative Ileus
Keywords: sham feeding; postoperative ileus; liver transplantation
MeSH Terms: interventions — Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- gum chewing (Experimental): Gum type was standardized with all subjects receiving sugar-free xylitol gum.
  The patients in the chewing gum group, gum chewing began the morning of postoperative day 1. Patients chewed gum (two tablets) 3 times daily in the morning, afternoon, and evening for 15 min. The administration of the therapy was implemented by ICU nurses and recorded in the clinical report form file. All gum-chewing patients completed their course of gum chewing until gas out.
  Interventions: Other: gum chewing
- Control (Placebo Comparator): Routine care during NPO
  Interventions: Other: Control

INTERVENTIONS:
Other: gum chewing — gum chewing
  Arms: gum chewing
Other: Control — Routine care during NPO
  Arms: Control

SUMMARY:
Postoperative ileus is a common after abdominal surgery. Multifactorial etiology such as surgical trauma, bowel manipulation and perioperative opioids contributes to delayed return of normal gut function Chewing gum has recently been used as a form of sham feeding to stimulate acceleration of gut function after abdominal surgery.

The investigators hypothesize that sham feeding with chewing gum will accelerate return of gut function after liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* elective liver transplantation surgery
* an ability to chew gum

Exclusion Criteria:

* emergency surgery
* age less than 18 years,
* inability to provide written informed consent
* an inability to chew gum
* hepaticojejunostomy
* sedated patients
* reintubated patients
* Glasgow Coma Scale <13
* reoperation before gas out
* previous bowel surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
time to flatus | an expected average of 75 hours

SECONDARY OUTCOMES:
percentage of target calories | an average 4 days
ICU length of stay | an average 96 hous
hospital length of stay | an average 20 days

CONTACTS AND LOCATIONS:
Overall Officials: Hogeol Ryu, MD. PhD., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea